CLINICAL TRIAL: NCT02294929
Title: Cryoballoon Ablation for Pulmonary Vein Isolation in Patients With Longstanding Persistent Atrial Fibrillation (the CRYO-LPAF Study)
Brief Title: Cryoballoon Ablation in Patients With Longstanding Persistent Atrial Fibrillation
Acronym: CRYO-LPAF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Uppsala University Hospital (Other)
Collaborators: Swedish Heart Lung Foundation (Other); Medtronic (Industry)
Responsible Party: Principal Investigator, Carina Blomstrom Lundqvist, Professor, Uppsala University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRYO-LPAF
Record Dates: First submitted 2014-11-12; First posted 2014-11-19 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Atrial Fibrillation
Keywords: catheter ablation; cryoballoon
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Atrial fibrillation ablation (Other): Cryoballoon ablation for pulmonary vein isolation
  Interventions: Procedure: Atrial fibrillation ablation

INTERVENTIONS:
Procedure: Atrial fibrillation ablation — Atrial fibrillation ablation using the Arctic Front™ Advance Cardiac CryoAblation Catheter in two balloon sizes (23mm and 28mm) for pulmonary vein isolation
  Other Names: Medtronic Arctic Front™ Advance Cardiac CryoAblation System; The Arctic Front™ Advance Cardiac CryoAblation Catheter; The FlexCath™ Steerable Sheath; CryoCath Cryoablation Console

SUMMARY:
Prospective and explorative clinical study. The objective is to assess the clinical efficacy of pulmonary vein isolation using the Arctic Front Advance cryoballoon in patients with longstanding persistent atrial fibrillation (AF) at one year follow up.

44 subjects will be enrolled. Patients with longstanding persistent AF, with continuous AF duration longer than one year, who have not previously undergone an AF ablation procedure, and have symptoms related to AF corresponding to at least European Heart Rhythm Association (EHRA) score 2, will be studied. Patients should have failed at least one betablocker or class I or III antiarrhythmic drug.

Excluded are those with congestive heart failure with New York Heart Association (NYHA) class 3 or more, left ventricular ejection fraction < 40%, left atrial diameter ≥ 60 mm, significant valvular disease or planned cardiac intervention within next 12 months, and conventional contraindications for AF ablation procedures.

Patients will be screened with echocardiography and response to electrical cardioversion. Following conversion to sinus rhythm, amiodarone will be initiated to maintain sinus rhythm. Pulmonary vein isolation will be performed using the Arctic Front Advance cryoballoon ablation catheter. Pulmonary vein conduction block will be assessed by a circular mapping catheter.

All patients will be subject to electroanatomical voltage mapping during sinus rhythm for demonstration of extent of atrial myocardial lesions after ablation.

Patients will be followed every third month up to one year after the ablation procedure. Arrhythmia monitoring during follow up will be performed by 7 day Holter monitoring at 6, 9 and 12 months follow up, including a 12 lead ECG. 12 months follow up for symptoms, EHRA score, and quality of life. Patients with symptomatic recurrence requiring a redo ablation procedure will be re-studied after 8-12 months while asymptomatic patients will be studied at 12 months follow up.

Primary end-Point is Clinical success based on symptoms and presence of AF. Secondary end-Points include freedom from AF without antiarrhythmic drugs at 6 and 12 months according to 7 day Holter and ECG, Rhythm, AF burden, AF profile, Quality of Life, Symptoms, Adverse Events, atrial size and function, Biomarkers, extent of scar tissue, predictive factors of freedom from AF, complications, hospitalization and Health economics.

DETAILED DESCRIPTION:
This is a prospective and explorative clinical study performed at one centre. Objective: The objective of this study is to assess the clinical efficacy of pulmonary vein isolation using the Arctic Front Advance cryoballoon in patients with longstanding persistent atrial fibrillation (AF) at one year follow up.

44 subjects will be enrolled. Clinical sites: Arrhythmia centre in Uppsala University Hospital, Uppsala Sweden.

Subject population: Patients with longstanding persistent AF, with continuous AF of longer duration than one year, who have not previously undergone an AF ablation procedure, and who have symptoms related to AF corresponding to at least EHRA score 2, will be studied. Atrial fibrillation should be confirmed on at least 2 consecutive ECG recordings during the past one year supporting the presence of AF for at least one year. Patients should have failed at least a betablocker or class I or III antiarrhythmic drug.

In order to exclude permanent AF patients, an electrical cardioversion with conversion to sinus rhythm maintained for at least one hour, is required.

Excluded patients are those with congestive heart failure with New York Heart Association (NYHA) class 3 or more, left ventricular ejection fraction (LVEF) < 40%, left atrial diameter (LA) ≥ 60 mm, significant valvular disease or planned cardiac intervention within the next 12 months, and conventional medical contraindications for AF ablation procedures.

Pulmonary vein isolation: Pulmonary vein isolation (PVI) will be performed using the Arctic Front Advance cryoballoon ablation catheter. Acute procedural success is defined as electrical isolation of all pulmonary veins assessed by entrance and exit block, including 20 minutes waiting time and the use of the provocative agent adenosine to screen for early recurrence of PV conduction.

Design of the study: Patients will be screened with echocardiography and response to electrical cardioversion. Following conversion to sinus rhythm, amiodarone will be initiated in order to maintain sinus rhythm.

After cryoballoon ablation of all pulmonary veins, PV conduction block will be assessed by a circular mapping catheter, including waiting time and provocative agents. All patients will be subject to electro anatomical voltage mapping during sinus rhythm for demonstration of the extent of atrial myocardial lesions after ablation. Biomarkers including nTproBNP and troponin I, reflecting myocardial strain and destruction, will be collected at baseline and at different time points after the procedure.

Patients will be followed every third month up to one year after the ablation procedure. Amiodarone will be withdrawn one month after the ablation procedure.

Arrhythmia monitoring during follow up will be performed by a 7 day Holter monitoring every third month at 6, 9 and 12 months follow up, including a 12 lead ECG.

A transthoracic echocardiography will be repeated at 12 months follow up to assess LA volume and contractility. Symptoms, EHRA score, and quality of life (QoL) will be evaluated. Predictive variables for successful outcome/AF recurrence will be analysed.

All patients will be reinvestigated for assessment of PV re-conduction using a circular mapping catheter, irrespective of symptoms. Patients with symptomatic recurrence requiring a redo ablation procedure will be re-studied after 8-12 months while asymptomatic patients will be studied at 12 months follow up.

Primary end-point:

Clinical success defined as

* Freedom from AF related symptoms, off or on previously ineffective antiarrhythmic drugs irrespective of the presence of asymptomatic AF on Holter. AF may be either absent or paroxysmal in nature, or
* Presence of AF related symptoms, off or on previously ineffective antiarrhythmic drugs, but with significant symptomatic improvement to the extent that a redo procedure or a novel previously not tested antiarrhythmic drug is not desired as declared by the patient on a symptom questionnaire. Atrial fibrillation may be either absent or paroxysmal as recorded on Holter or ECG tracings after 1 or 2 procedures at 12 months.

Secondary end-points:

1. Complete freedom from AF without antiarrhythmic drugs at 6 and 12 months after 1-2 ablation procedures according to 7 day Holter and ECG.
2. Rhythm (% of subjects in sinus rhythm, paroxysmal AF and persistent AF) at 12 months.
3. AF burden on 7 day Holter at 12 months.
4. AF profile
5. Assess whether PVI is crucial for elimination of AF in patients with longstanding persistent AF. Correlation between freedom from AF/recurrence and PV isolation/re-conduction at repeat electrophysiological study.
6. Systemic blood pressure.
7. Quality of Life determined by standardized questionnaires (SF 36, with all domains and time-points and EQ 5D).
8. Symptoms (Symptoms Severity Questionnaire and EHRA Symptom Classification).
9. Incidence, intensity and relationship of Adverse Events.
10. Left and right atrial size and function (sinus rhythm) (echocardiography corrected for Body Surface area, dPdT) prior to and after ablation at 12 months.
11. Biomarkers including nTproBNP and troponin I, reflecting myocardial strain and destruction, will be collected at baseline and at different time points after the procedure. A biomarker reflecting fibrosis and brain damage will be analysed.
12. Extent of scar tissue as indicated by LA voltage mapping at baseline and extent of electrical silence around PV postablation.
13. A subgroup analysis will determine whether sinus rhythm obtained by AF ablation is superior AF with regard to all secondary endpoints including QoL, Symptoms, cardiovascular hospitalizations, safety, biomarkers, left atrial size and function, at 12 months.
14. Prediction of freedom from AF by risk variables including LA volume, LA contractility (strain rate), LA intracardiac pressures and dpdt, Atrial amplitude analysis during AF prior ablation, extent of scar tissue as assessed by a voltage mapping at baseline during sinus rhythm, biomarkers, and demographic variables (AF duration, hypertension, ischemic heart disease, diabetes and CHADS2VASscore).
15. Catheter related complications.
16. Cardiovascular hospitalization
17. Health economics

ELIGIBILITY:
Inclusion Criteria:

1. Patients with longstanding persistent AF, with continuous AF of greater than one year, as verified by ECG or telemetry strip at least one year ago, and at inclusion but with no documentation of sinus rhythm in between.
2. Atrial fibrillation should be confirmed on at least 2 consecutive ECG supporting the presence of AF for at least one year.
3. Patients with symptoms corresponding to at least EHRA score 2.
4. Patients, who have not previously undergone an AF ablation procedure, should have failed at least a betablocker or class I or III antiarrhythmic drug.

Exclusion Criteria:

1. Sinus rhythm cannot be maintained for at least 1 minute after an electrical cardioversion.
2. Congestive heart failure with NYHA class 3 or more.
3. LVEF < 35% which is not secondary to AF with inadequate rate control, according to the judgement of the investigator.
4. LA diameter ≥ 55 mm by echocardiography.
5. Prior AF ablation procedure of any kind.
6. AF secondary to a transient or correctable abnormality including electrolyte imbalance, trauma, recent surgery, infection, toxic ingestion, and uncontrolled thyroid disease as well as AF triggered by other uniform supraventricular tachycardia.
7. Contraindication to treatment with Warfarin or other anticoagulants.
8. Significant valvular disease or planned cardiac intervention.
9. Hypertrophic cardiomyopathy.
10. Recent cardiac disease states within the last 6 months; unstable angina, acute myocardial infarction, revascularisation procedures, valve disease
11. Implantable cardioverter-defibrillator (ICD), biventricular pacing device, or Dual chamber- or single chamber pacemaker patients who are dependent on ventricular pacing
12. Patients with intra-atrial thrombus, tumor, pulmonary embolism or another abnormality in whom transseptal catheterization or appropriate vascular access is precluded.
13. Renal failure requiring dialysis or abnormalities of liver function tests.
14. Participant in investigational clinical or device trial.
15. Unwilling or unable to give informed consent or inaccessible for follow-up and psychological problem that might limit compliance.
16. Active abuse of alcohol or other substance which may be causative of AF and/or might affect compliance.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-09 (Actual); Primary Completion 2018-09 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Clinical success | 12 months
  Clinical success defined as:
  * Freedom from AF related symptoms, off or on previously ineffective antiarrhythmic drugs irrespective of the presence of asymptomatic AF on Holter provided AF is absent or paroxysmal in nature AF, or
  * Presence of AF related symptoms, off or on previously ineffective antiarrhythmic drugs, but significant symptomatic improvement to the extent that a redo procedure or a novel previously not tested antiarrhythmic drug is not desired as declared by the patient on a symptom questionnaire. Atrial fibrillation may be either absent or paroxysmal as recorded on Holter or ECG tracings after 1 or 2 procedures at 12 months.

SECONDARY OUTCOMES:
Complete freedom from AF | 6, 12 months
  Complete freedom from AF without antiarrhythmic drugs after 1-2 ablation procedures according to 7 day Holter and ECG
Rhythm assessed by % of subjects in sinus rhythm, paroxysmal AF and persistent AF | 12 months
  % of subjects in sinus rhythm, paroxysmal AF and persistent AF
Atrial Fibrillation burden | 12 months
  AF burden on 7 day Holter defined as time spent in AF as recorded by Holter monitoring
Role of Pulmonary vein isolation for elimination of atrial fibrillation | 12 months
  Correlation between AF recurrence and re-conduction at repeat EP study.
Quality of life | 12 months
  Quality of Life (Short form (SF)-36 all domains and time-points.
Symptoms Severity Questionnaire and EHRA Symptom Classification | 12 months
  Symptom Severity Questionnaire and EHRA Symptom Classification
Biomarkers | Baseline, 6 hours, 24 hours, 12 months
  Biomarkers reflecting myocardial strain and destruction (Troponin I, Nt-proBNP), collected at baseline and at different time points after the procedure. A biomarker reflecting fibrosis (TGF-β1 and aminoterminal peptide of procollagen type III) and brain damage (S100β, a dimeric calcium-binding protein) will be analysed.
Scar tissue | 12 months
  Extent of scar tissue as indicated by left atrial voltage mapping at baseline and extent of electrical silence around pulmonary vein postablation, and measures of intra-atrial conduction times in right and left Atria.
Prediction of freedom from AF | 12 months
  Prediction of freedom from AF by risk variables including left atrial (LA) volume, LA contractility, intracardiac pressures and LA dPdT, Atrial amplitude analysis during AF prior ablation, extent of scar tissue as assessed by a voltage mapping, biomarkers and demographic variables variables (AF duration, hypertension, ischemic heart disease, diabetes and CHADS2VASscore)
Health economics | 12 months
  Quality of Life assessed by EuroQual (EQ) 5D and all Cardiovascular hospitalizations, interventions and events.
Catheter related complications | 12 months
  Catheter related complications at and after ablation
Left and right atrial size and function | 12 months
  Left and right atrial size and function (sinus rhythm) (echocardiography corrected for body Surface area)

OTHER OUTCOMES:
Is sinus rhythm obtained by AF ablation superior to AF with regard to all secondary endpoints ? | 12 months
  Determine whether sinus rhythm obtained by AF ablation is superior to AF with regard to all secondary endpoints including QoL, Symptoms, cardiovascular hospitalizations, safety, biomarkers, left atrial size and function.

CONTACTS AND LOCATIONS:
Overall Officials: Carina M Blomström Lundqvist, Professor, Principal Investigator — Department of Cardiology, Uppsala University Hospital
Locations (1):
- Carina Blomström Lundqvist, Uppsala, Sweden

REFERENCES:
- [Result] Aytemir K, Gurses KM, Yalcin MU, Kocyigit D, Dural M, Evranos B, Yorgun H, Ates AH, Sahiner ML, Kaya EB, Oto MA. Safety and efficacy outcomes in patients undergoing pulmonary vein isolation with second-generation cryoballoondagger. Europace. 2015 Mar;17(3):379-87. doi: 10.1093/europace/euu273. Epub 2014 Nov 5. PMID 25376699